CLINICAL TRIAL: NCT03571555
Title: A Prospective Cohort Study Evaluating a Psychosocial Programme for Adolescents Living With HIV and Their Caregivers in Botswana
Brief Title: Prospective Cohort Study of Adolescents Living With HIV and Their Caregivers Attending a Psychosocial Programme in Botswana
Status: Completed | Type: Observational
Sponsor: Royal Holloway University (Other)
Collaborators: African Comprehensive HIV/AIDS Partnership (Other); Sentebale (Other)
Responsible Party: Principal Investigator, Dr. Michael Evangeli, Principal Investigator, Royal Holloway University
Other Study IDs: Sentebale
Record Dates: First submitted 2018-05-31; First posted 2018-06-27 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Hiv
Keywords: HIV; perinatal; adolescent; camp; psychosocial
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Muscle Cramp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young people with perinatally acquired HIV: Residential interventions (camps) and community based support (clubs)
  Interventions: Behavioral: Sentebale Psychosocial Programme
- Caregivers of young people with perinatally acquired HIV: Community based support (clubs)
  Interventions: Behavioral: Sentebale Psychosocial Programme

INTERVENTIONS:
Behavioral: Sentebale Psychosocial Programme — Residential interventions (camps) for the young people, and community based support (clubs) for the young people and the caregivers.

SUMMARY:
Adolescents/young adults with perinatally acquired HIV (PAH) face a number of antiretroviral (ART) adherence and well-being challenges. Two psychosocial interventions that have been developed to address a range of needs of this population (and their caregivers) are residential interventions (camps) and support groups (clubs). There has been little quantitative evaluation of the effects of attending camps for young people and clubs (for children or caregivers), globally. This study aims to investigate whether a package of psychosocial support (camps and clubs) offered to young people living with HIV and their caregivers in Botswana by the Sentebale organisation, is associated with improvements in psychological, behavioural and clinical outcomes from first attendance to one year follow-up. In addition, the study will explore how the psychosocial programme is experienced by young people and their caregivers, and what the perceived impact is. The project as a whole will take place over three years. There will be an initial six month preparatory phase that will include the adaptation of self-report measures for the study context. Subsequently, two studies will be undertaken. The main study will involve a single group within-participants prospective cohort design with two time points (baseline and one year follow-up) with young people and caregivers. The sub-study will involve a qualitative cross sectional design involving semi-structured interviews with young people and caregivers. Young people will be eligible to participate if they are aged 10 to 19 years at the time of study enrolment, are living with HIV and aware of HIV-positive status, have recently started attending the Sentebale programme, and are able to give informed assent/consent. We will aim to retain 175 young people (of 253 recruited) . We will also aim to retain 178 caregivers (of 263 recruited). The sample size for the sub-study will consist of ten young people and ten caregivers.

DETAILED DESCRIPTION:
There are approximately two million young people between 10 and 19 years, living with HIV (UNAIDS, 2013). Many of this population have been living with HIV since birth. Adolescents/young adults with perinatally acquired HIV (PAH) face a number of antiretroviral (ART) adherence and well-being challenges. They often have long histories of ART use with suboptimal regimens (Sohn & Hazra, 2013) and rates of viral suppression are variable, often associated with poor ART adherence (Kim, Gerver, Fidler, & Ward, 2014). Challenges to positive well-being in young people with PAH include some experiencing multiple caretaking transitions, loss due to parental illness or death, and other stressors associated with living with a chronic and stigmatised illness (e.g., hospitalisations, missed school and social opportunities, HIV disclosure challenges and pain). There is evidence of lower levels of wellbeing in young people living with PAH compared to their HIV unaffected peers (Mellins & Malee, 2013).

Offering psychosocial interventions for young people living with HIV has the potential for enhancing well-being, HIV adjustment, ART adherence, self-esteem and increasing HIV knowledge and HIV disclosure. There are a small number of quantitative studies evaluating interventions to enhance antiretroviral adherence in young people with HIV (Shaw & Amico, 2016) but few robust quantitative evaluations of psychosocial interventions to enhance well-being in this population (King, De Silva, Stein, & Patel, 2009). There are no interventions on enhancing onward HIV disclosure in adolescents living with HIV (Evangeli & Foster, 2014).

Two psychosocial interventions that have been developed to address a range of needs of this population (and their caregivers) are residential interventions and support groups. Regarding residential interventions, there is quantitative evidence in other chronic conditions of increased youth self-esteem after attendance (Odar, Canter, & Roberts, 2013). There is also some qualitative literature on evaluating residential interventions (support camps) for young people living with HIV in the US (Gillard & Allsop, 2016; Gillard, Witt, & Watts, 2011; Pearson, Johnson, Simpson, & Gallagher, 1997). Interviews with Camp attendees have revealed that this intervention can elicit a sense of belonging, enjoyment, escape, personal growth, being oneself, and caring connections, as well as increasing HIV knowledge, attitudes and skills. A recent quantitative evaluation of a residential intervention in the UK showed evidence for increases in HIV knowledge and pro-HIV disclosure attitudes and cognitions that were maintained at six month follow-up (Evangeli, Lut, & Ely, 2016).

There is also some global evidence of positive benefits of support groups for children living with HIV, who report that groups provide a sense of belonging, normality, confidence and safety; supportive relationships; and a place to learn about treatment adherence and living healthily (Brothers, Harper, Fernandez, Hosek, & Adolescent Trials Network for, 2014; Funck-Brentano et al., 2005; Midtbo, Shirima, Skovdal, & Daniel, 2012; Mupambireyi, Bernays, Bwakura-Dangarembizi, & Cowan, 2014; Muskat, Salter, Shindler, Porter, & Bitnum, 2016). There has been little quantitative evaluation of the effects of attending support groups (for children or caregivers), although one pilot study using non-random allocation, showed some evidence of decreased worry about illness, less negative perception about treatment and greater rates of viral suppression in adolescents living with HIV (Funck-Brentano et al., 2005).

Sentebale is an organisation that has been providing residential interventions (camps) to adolescents living with HIV, and follow up support groups (clubs) for these adolescents and their caregivers, amongst other psychosocial interventions, in Lesotho for a number of years. Sentebale is now offering a similar package of psychosocial services to young people and caregivers in Botswana, partnering with Serious Fun Children's Network. The aims of Sentebale are to provide support that will enable young people to living healthy and hopeful lives, increase confidence, improve educational and occupational functioning, increase care and support, enhance HIV communication, increase caregiver support, reduce onward transmission, and increase remembering to take medication. We will evaluate the above psychosocial programme, given the need to investigate the psychosocial, behavioural and clinical outcomes of this type of intervention in high HIV prevalence contexts. Botswana has an estimated HIV prevalence of 6.6% in 15-19 year olds, and an estimated adult prevalence rate of 18.5%, and despite high levels of ART adherence, psychological difficulties in this population are common (Gupta et al., 2010).

Aims and objectives

This three year study aims to answer the following questions in a population of adolescents living with HIV and their caregivers:

1. Is the package of support offered by Sentebale (camps for young people, clubs for young people and caregivers) associated with improvements in psychological, behavioural and clinical outcomes from first attendance to one year follow-up?
2. How is the package of support experienced by young people and their caregivers, and what is the perceived impact for young people and their caregivers?

Study Design

1. Main study - single group within-participants prospective cohort design with two time points (baseline and one year follow-up) with 175 young people and 178 caregivers retained in the study (Study Aim 1).
2. Sub-study - qualitative cross sectional design involving semi-structured interviews with 10 young people and 10 caregivers (Study Aim 2).

ELIGIBILITY:
YOUNG PEOPLE

Inclusion Criteria:

* Aged 10 to 19 years at the time of study enrolment
* Living with HIV and aware of HIV-positive status
* Able to give informed consent if 18 or 19 years
* Able to give informed assent if 10-17 years
* Presence of a caregiver to give caregiver consent if 10-17 years
* Attending Sentebale clubs with first attendance at club within previous month

Exclusion Criteria:

* Previous camp attendance
* Any attendance at a different club/organisation providing a similar function
* Planning to leave the area served by the club within the next year

CAREGIVERS

Inclusion Criteria:

* Primary caregiver for a young person attending Sentebale
* Able to give informed consent
* Attending Sentebale clubs with first attendance within previous month

Exclusion Criteria

* Any attendance at a different club/organisation providing a similar function
* Planning to leave the area served by the club within the next year

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 10-19 year olds living with HIV, new attenders to the Sentebale psychosocial programme
  Primary caregivers of 10-19 year olds living with HIV attending Sentebale, who are also attending Sentebale themselves
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sentebale, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: Yes
Anonymised electronic data from the study will be transferred to a data repository (eg.,Figshare or RHUL Research Data Archive) at the end of the study.
Supporting Information: Study Protocol
Time Frame: At the end of the study. For 10 years.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not assigned to groups. The study was an uncontrolled cohort study.
Period: Overall Study
Arm/Group | Young People With Perinatally Acquired HIV | Caregivers of Young People With Perinatally Acquired HIV
Started | 252 | 263
Completed | 177 | 195
Not Completed | 75 | 68

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Young People With Perinatally Acquired HIV | Caregivers of Young People With Perinatally Acquired HIV | Total
Number analyzed (Participants) | 252 | 263 | 515
Age, Customized [Median (Inter-Quartile Range); unit: years] | 16 [14 to 17] | 43 [38 to 48] | 30 [18 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 242 | 371
  Male | 123 | 21 | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Botswana | 252 | 263 | 515

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life/Well-being (Young People)
Description: The 17 item Pediatric Symptom Checklist (PSY-Y-17) will be used.
  Minimum value 0, maximum 51. Higher scores, worse outcome.
Time Frame: One year
Population: Young people with perinatally acquired HIV
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Young People With Perinatally Acquired HIV | Caregivers of Young People With Perinatally Acquired HIV
Number analyzed (Participants) | 249 | 0
score on a scale | 4.77 (4.21) |

2. Secondary Outcome: HIV Knowledge (Young People)
Description: The Brief HIV Knowledge Questionnaire (Carey & Schroder, 2002) and other measures (Aaro et al, 2011; Evangeli et al, 2016) will be adapted to produce a new measure of general HIV knowledge, transmission, medication and reproduction information.
Time Frame: One year
Reporting Status: Not Posted

3. Secondary Outcome: HIV Adjustment (Young People)
Description: The 18 item Illness Cognition Questionnaire will be used (Evers et al., 2001).
Time Frame: One year
Reporting Status: Not Posted

4. Secondary Outcome: ART Adherence Behaviour (Young People)
Description: The total score of the CASE adherence index (Mannheimer et al., 2006) will be used. Higher scores indicate higher self-reported ART adherence
Time Frame: One year
Reporting Status: Not Posted

5. Secondary Outcome: ART Adherence Attitudes (Young People)
Description: The total score of 15 item antiretroviral medication attitudes scale (Viswanathan, Anderson, & Thomas, 2005) will be used. Higher scores indicate more positive adherence attitudes.
Time Frame: One year
Reporting Status: Not Posted

6. Secondary Outcome: ART Adherence Self-efficacy (Young People)
Description: The total score of the 12 item HIV medication self-efficacy scale (Erlen, Cha, Kim, Caruthers, & Sereika, 2010) will be used. Higher scores indicated higher adherence self-efficacy.
Time Frame: One year
Reporting Status: Not Posted

7. Secondary Outcome: HIV Onward Disclosure Cognitions and Affect (Young People)
Description: The 18 item Adolescent HIV Disclosure Cognitions and Affect Scale (Evangeli, 2017) will be used to assess attitudes towards sharing one's status, normative disclosure beliefs, disclosure affect and disclosure self-efficacy.
Time Frame: One year
Reporting Status: Not Posted

8. Secondary Outcome: HIV Onward Disclosure (Young People)
Description: The 18 item Adolescent HIV Disclosure Cognitions and Affect Scale (Evangeli, 2017) will be used to assess attitudes towards sharing one's status, normative disclosure beliefs, disclosure affect and disclosure self-efficacy. The total score will be used. Higher scores indicate more pro-disclosure beliefs. An additional item assessed the young person's intention to share their status with others over the next year will be added.
  HIV disclosure events will be assessed at baseline and follow-up through recording the frequency of new disclosures in last year (first hand or second hand) and the proportion in one's social network disclosed to (Serovich, Craft, & Reed, 2012; Serovich, Craft, & Yoon, 2007).
Time Frame: One year
Reporting Status: Not Posted

9. Secondary Outcome: HIV Onward Disclosure Behaviour (Young People)
Description: HIV disclosure events will be assessed at baseline and follow-up through recording the frequency of new disclosures in last year (first hand or second hand) and the proportion in one's social network disclosed to (Serovich, Craft, & Reed, 2012; Serovich, Craft, & Yoon, 2007).
Time Frame: One year
Reporting Status: Not Posted

10. Secondary Outcome: HIV Communication Behaviour (Young People)
Description: The frequency of HIV communication will be measured.
Time Frame: One year
Reporting Status: Not Posted

11. Secondary Outcome: HIV Communication Beliefs (Young People)
Description: The Adolescent HIV Communication Belief Scale (Evangeli, in press) will be used. An additional item will assess intention to communicate about HIV.
Time Frame: One year
Reporting Status: Not Posted

12. Secondary Outcome: Self-esteem (Young People)
Description: The 10 item Rosenberg global self-esteem measure will be used (Rosenberg, 1965).
Time Frame: One year
Reporting Status: Not Posted

13. Secondary Outcome: HIV Stigma (Young People)
Description: The total score of the 10 item Stigma Scale - Revised (Wright, Naar-King, Lam, Templin, & Frey, 2007) will be used. Higher scores indicate more HIV stigma
Time Frame: One year
Reporting Status: Not Posted

14. Secondary Outcome: Social Support (Young People)
Description: The total score of the 11 item Child and Adolescent Social Support Scale (Malecki & Demaray, 2002) will be used. Higher scores indicate greater social support
Time Frame: One year
Reporting Status: Not Posted

15. Secondary Outcome: Hope(Young People)
Description: The total score of the 5 item Botswana Adolescent Beliefs about the Future Scale will be used. Higher scores indicate greater hope.
Time Frame: One year
Reporting Status: Not Posted

16. Secondary Outcome: HIV Knowledge (Caregivers)
Description: The HIV-KQ-18 measure (Carey & Schroder, 2002) will be adapted for use in Botswana
Time Frame: One year
Reporting Status: Not Posted

17. Secondary Outcome: ART Adherence Attitudes (Caregivers)
Description: The 15 item antiretroviral medication attitudes scale (Viswanathan et al., 2005) will be used. The measure will be adapted for use with Batswana caregivers.
Time Frame: One year
Reporting Status: Not Posted

18. Secondary Outcome: HIV Stigma (Caregivers)
Description: The total score of the 9 item HIV Stigma Scale will be used (Kalichman et al., 2005). Higher scores indicate higher levels of HIV stigma.
Time Frame: One year
Reporting Status: Not Posted

19. Secondary Outcome: Viral Suppression (Young People)
Description: Most recent viral load in the six months before the baseline assessment and most recent viral load in the six months after the follow-up period, will be collected from participants' clinical records.
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | Young People With Perinatally Acquired HIV | Caregivers of Young People With Perinatally Acquired HIV
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/263
Serious Adverse Events (participants affected / at risk) | 0/252 | 0/263
Other Adverse Events (participants affected / at risk) | 0/252 | 0/263

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT03571555/Prot_SAP_000.pdf